CLINICAL TRIAL: NCT06254768
Title: Use of Continuous Glucose Monitors in Children and Adolescents With Obesity
Acronym: CGM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Sri Nikhita Chimatapu, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 22-000958
Record Dates: First submitted 2023-02-27; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Unblinded (Experimental): They will wear the device and have access to their data- UNBLINDED ARM
  Interventions: Device: Continuous glucose monitor
- Blinded (Experimental): They will wear the device but will not have access to their data- BLINDED ARM
  Interventions: Device: Continuous glucose monitor

INTERVENTIONS:
Device: Continuous glucose monitor — its a device used to measure glucose from interstitial fluids and provides feedback regarding the same every 5 minutes.

SUMMARY:
To study if continuous glucose monitors are feasible for use in children and adolescents with obesity.

DETAILED DESCRIPTION:
Various CGMs are approved by the U.S. Food and Drug Administration (FDA) for use in children and adults with diabetes. However, to date, little is known about how CGM technology can be integrated into weight management strategies for adolescents with obesity. No study to date has explored the effects of unblinded vs. blinded CGM use alone, without any other lifestyle modification recommendations. Thus, to address this question, this is a cross-over feasibility trial of blinded vs. unblinded CGM use in youth with obesity. This study hypothesizes that CGM will be a feasible and acceptable technology for youth with obesity, without diabetes, to utilize, and that access to daily glucose trends will facilitate positive changes in eating behavior and daily activity level compared to blinded CGM use. Thirty adolescents with obesity will be recruited into a six-week cross-over trial. All participants will be randomly assigned to either the blinded or unblinded group for three weeks. And then cross over to the other group for another three weeks. The primary endpoints are recruitment, retention, and adherence. While the secondary endpoints are glycemic variability, as captured on CGM, change in weight as an excess percentage of 95th percentile, sleep, dietary intake, physical activity, and eating behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-21 years BMI >95th percentile

Exclusion Criteria:

* Previous diagnosis of Prader Willi Syndrome or hypothalamic obesity
* Intellectual disability
* Previous or planned bariatric surgery
* Hemoglobin A1c >6.5 %
* Current use of medication that impacts weight

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of continuous glucose monitor(CGM) use in children and adolescents with obesity | 6 weeks
  Investigator will measure this outcome using recruitment rate achieved each month for the duration of the study period as the number of participants screened per month over the number of participants consented.

SECONDARY OUTCOMES:
To access the change in glycemic variability measured by CGMS in unblinded versus blinded periods through standard deviation of the mean. | 6 weeks
  Investigator will measure the effect of un-blinded CGM versus blinded use on glycemic variability measured by the Standard Deviation of the mean glycemia (SD) measured by CGMS.

OTHER OUTCOMES:
Effect of on sleep in youth with obesity using CGMs | 6 weeks
  Investigator will assess the effect on quality of sleep in youth with obesity when using CGMs with the help of Pittsburgh Sleep Quality Index. The Pittsburgh Sleep Quality Index scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Effect of CGM use on physical activity in youth with obesity when using CGMs | 6 weeks
  Investigator will assess the effect on physical activity when using CGMS with the help of International Physical Activity Questionnaire. The items on the form are structured to provide separate scores on walking, moderate-intensity and vigorous-intensity activity. Computation of the total score for the short form requires summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activities.
Effect of CGM use on dietary intake in youth with obesity when using CGMs | 6 weeks
  Investigator will assess the effect on dietary intake when using CGMS with the help of The Automated Self-Administered 24-hour Dietary Assessment Tool which is a tool that enables multiple, automatically coded, self-administered 24-hour diet recalls and/or single or multi-day food records, also known as food diaries.
Effect of CGM use on eating behaviors in youth with obesity when using CGMs | 6 weeks
  Investigator will assess the effect on eating behaviors in youth with obesity when using CGMs with the help of Dutch Eating Behavior Questionnaire. Items on the Dutch Eating Behavior Questionnaire range from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behavior.
Effect of CGM use on change in the BMI as a percentage of the 95th percentile (%BMIp95) in youth with obesity when using CGMs | 6 weeks.
  Investigator will measure the change in the BMI as a percentage of the 95th percentile (%BMIp95) in youth with obesity when using CGMs between baseline to week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Mittelman, MD, PhD, Study Director — University of California, Los Angeles
Locations (1):
- Pediatric Endocrinology Division, University of California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No